CLINICAL TRIAL: NCT02645799
Title: Biorest Liposomal Alendronate Administration for Diabetic Patients Undergoing Drug-Eluting Stent Percutaneous Coronary Intervention
Brief Title: BLADE-PCI Trial (BLADE); PHASE IIB LIPOSOMAL ALENDRONATE STUDY
Acronym: BLADE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BIOrest Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LA-II-02
Record Dates: First submitted 2015-12-24; First posted 2016-01-05 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LABR-312 (Active Comparator): LABR-312 will be administered intravenously at the time of percutaneous coronary intervention (PCI) with a drug eluting stent. Target lesions will be treated with the Resolute Integrity Drug Eluting Stent during the index PCI.
  Three (3) doses will be tested:
  Group 1: Low dose -> 0.01 mg LABR-312 Group 2: Intermediate dose-> Up to 0.03 mg LABR-312 Group 3: High dose-> Up to 0.08 mg LABR-312 The duration of subject participation will be 1 year; clinical follow-up will be performed at 30 days, 9 months, and 1 year post randomization.
  OCT follow-up will be performed at 9 months.
  Interventions: Drug: LABR-312
- saline (Placebo Comparator): Placebo will be administered intravenously at the time of percutaneous coronary intervention (PCI) with a drug eluting stent. Target lesions will be treated with the Resolute Integrity Drug Eluting Stent during the index PCI.
  Three (3) doses will be tested:
  Group 1: Low dose -> placebo (saline) equivalent to 0.01 mg LABR-312. Group 2: Intermediate dose-> placebo (saline) equivalent to up to 0.03 mg LABR-312 Group 3: High dose-> placebo (saline) equivalent to up to 0.08 mg LABR-312. The duration of subject participation will be 1 year; clinical follow-up will be performed at 30 days, 9 months, and 1 year post randomization.
  OCT follow-up will be performed at 9 months.
  Interventions: Drug: Saline (placebo)

INTERVENTIONS:
Drug: LABR-312 — administered intravenously at the time of percutaneous coronary intervention (PCI) with a drug eluting stent
  Arms: LABR-312
Drug: Saline (placebo) — administered intravenously at the time of percutaneous coronary intervention (PCI) with a drug eluting stent
  Arms: saline

SUMMARY:
The main objective of this study is to assess the safety, efficacy and dose response of LABR-312 administered intravenously at the time of percutaneous coronary intervention (PCI) with a drug eluting stent in reducing restenosis as measured by Optical Coherence Tomography (OCT) at 9 months post procedure in patients with diabetes mellitus (DM).

Administration of LABR-312 at the time of PCI will reduce restenosis compared with placebo as assessed by the OCT endpoint of % neointimal hyperplasia (%NIH) volume at 9 months in patients with DM.

DETAILED DESCRIPTION:
This is a phase IIb, prospective, multi-center, multi-national, randomized, double-blind, two-arm, 1:1 (escalating dose LABR-312 vs. placebo) clinical trial.

In both study arms, all target lesions will be treated with the Resolute Integrity Drug Eluting Stent during the index PCI.

Lesions that are planned to be treated must be declared and recorded at the time of randomization.

Randomization will be stratified by the presence or absence of insulin treatment, HbA1c level (<7.5% vs. ≥7.5%), and by pre-procedure monocyte count (≥500/uL or below).

Subjects (n=~270) will be randomized to receive either the study drug LABR-312 or the placebo. Conditionally to ongoing safety monitoring, dose escalation of LABR-312 in the study arm will be performed: 0.01 mg (first 45 patients vs. 45 patients receiving placebo), up to 0.03 mg (next consecutive 45 patients vs. 45 patients receiving placebo) and up to 0.08 mg (final 45 consecutive patients vs. 45 patients receiving placebo). If a decision is made not to dose escalate, recruitment will continue with the highest dose level deemed safe by the ongoing safety monitoring, until approximately 270 subjects are randomized.

In the LABR-312 group, 3 doses will therefore be tested, resulting in 6 possibilities:

Group 1: Low dose 0.01 mg LABR-312 or equivalent volume of placebo (saline) administered IV.

Group 2: Intermediate dose Up to 0.03 mg LABR-312 or equivalent volume of placebo (saline) administered IV.

Group 3: High dose Up to 0.08 mg LABR-312 or equivalent volume of placebo (saline) administered IV.

The duration of subject participation will be 1 year; clinical follow-up will be performed at 30 days, 9 months, and 1year post randomization.

OCT follow-up will be performed at 9 months.

ELIGIBILITY:
General Inclusion Criteria: all must be present

1. Patient has medically treated diabetes mellitus (is on insulin or oral or injectable hypoglycemic medications).
2. Patient is eligible and has an indication for PCI with a drug eluting stent (patient may be consented prior to diagnostic angiography with possible PCI).
3. Patient presents with angina (stable or unstable), silent ischemia (in absence of symptoms must have a positive stress test, FFR ≤0.80, or angiographic stenosis of ≥70%), NSTEMI, or recent STEMI (>7 days from procedure).
4. Non-target vessel PCI are allowed prior to randomization depending on the time interval and conditions as follows:

   * During Baseline Procedure:
   * PCI of non-target vessels performed during the baseline procedure itself immediately prior to randomization, if successful and uncomplicated, defined as: <50% visually estimated residual diameter stenosis, TIMI Grade 3 flow, no dissection ≥ NHLBI type C, no perforation, no persistent ST segment changes, no prolonged chest pain, no TIMI major or BARC type 3 bleeding.

     * Less than 24 hours prior to Baseline Procedure:
   * Not allowed (see exclusion criteria #2).

     * 24 hours-30 days prior to Baseline Procedure:
   * PCI of non-target vessels 24 hours to 30 days prior to randomization if successful and uncomplicated as defined above.
   * In cases where non-target lesion PCI has occurred 24-72 hours prior to the baseline procedure, at least 2 sets of cardiac biomarkers must be drawn at least 6 and 12 hours after the non-target vessel PCI.
   * If cardiac biomarkers are initially elevated above the local laboratory upper limit of normal, serial measurements must demonstrate that the biomarkers are falling.

     * Over 30 days prior to Baseline Procedure:
   * PCI of non-target vessels performed greater than 30 days prior to procedure whether or not successful and uncomplicated.
5. All non-target lesions (i.e. those not meeting angiographic criteria for the study) should be treated prior to randomization. All target lesions must be planned to be treated during the index procedure. The investigator will declare which target lesions are intended for treatment at the time of randomization. In the event that all target lesions cannot be treated (e.g. due to contrast load), staged procedure should be delayed preferably at least 2 weeks after the index PCI, and those lesions will be considered non-target lesions. Any such planned staged lesions must be declared at the end of the index procedure.
6. Prior target-vessel PCI is allowed if it occurred ≥6 months prior to randomization and no restenosis is present, or if re-intervention is planned on the restenotic lesion(s) as a non-target lesion.
7. The patient or legal guardian is willing and able to provide written informed consent and comply with follow-up visits and the testing schedule.

Angiographic Inclusion Criteria (visual estimate) (all must be present):

1. Target lesion(s) must be located in a native coronary artery with visually estimated diameter of ≥2.25mm to ≤4.2mm and diameter stenosis ≥50% to <100%.
2. Thrombolysis in Myocardial Infarction (TIMI) flow 2 or 3. If more than 1 target lesion will be treated, the reference vessel diameter and lesion length of each must meet the above criteria.

General Exclusion Criteria: all must be absent

1. STEMI within 7 days of presentation to the first treating hospital, whether a transfer facility or the study hospital
2. PCI within the 24 hours prior to randomization
3. Cardiogenic shock (defined as persistent hypotension [systolic blood pressure <90 mm Hg] or requiring pressors or hemodynamic support, including IABP)
4. Known left ventricular ejection fraction <30%
5. Relative or absolute contraindication to DAPT for 6 months (including planned surgeries that cannot be delayed or chronic oral anticoagulant requirement, such as atrial fibrillation or prosthetic heart valve)
6. Hemoglobin <10 g/dL
7. Platelet count <100,000 cells/mm3 or >700,000 cells/mm3
8. White blood cell count <3,000 cells/mm3
9. Major and clinically significant active infection
10. Clinically significant liver disease
11. Renal insufficiency as defined by an estimated Glomerular Filtration Rate, GFR <40 ml/min by the MDRD formula
12. Active peptic ulcer or active bleeding from any site
13. Bleeding from any site requiring active medical attention within the prior 8 weeks
14. History of bleeding diathesis or coagulopathy or likely to refuse blood transfusions
15. Cerebrovascular accident (CVA) or has any permanent neurological defect as a result of CVA
16. Known allergy to the study stent components or protocol-required concomitant medications: alendronate, liposomal medications, aspirin, clopidogrel and prasugrel and ticagrelor, heparin and bivalirudin, or iodinated contrast that cannot be adequately pre-medicated
17. Subject is taking Bisphosphonates, including Alendronate (Fosamax); Clodronate (Bonefos); Etidronate (Didronel / Didrocal); Ibandronate (Bondronat); Pamidronate (Aredia); Risedronate (Actonel); Tiludronate (Skelid); Zoledronic acid (Zometa), or any other bisphosphonates not listed above.
18. Any co-morbid condition that may cause non-compliance with the protocol (e.g. dementia, substance abuse, etc.) or reduce life expectancy to <24 months (e.g. cancer, heart failure, lung disease)
19. Patient is participating in or plans to participate in any other investigational drug or device trial that has not reached its primary endpoint.
20. Women who are pregnant or breastfeeding (women of child-bearing potential must have a negative pregnancy test within one week before index procedure).
21. Women who intend to become pregnant within 12 months after the index procedure
22. Patient has received an organ transplant or is on a waiting list for an organ transplant.
23. Patient is receiving or scheduled to receive chemotherapy within 30 days before or any time after the index procedure.
24. Patient is receiving oral or intravenous immunosuppressive therapy or has known life-limiting immunosuppressive or autoimmune disease. Inhaled steroid and steroid use for contrast-allergy prophylaxis or treatment are allowed.

Angiographic Exclusion Criteria (visual estimate) (all must be absent):

1. Unprotected left main lesions >30% or left main intervention.
2. Primary PCI for STEMIOstial RCA lesion within 5 mm of ostium*
3. Coronary artery disease judged more suitable for surgical revascularization per guidelines and local heart team discussion.
4. Another lesion in either the target vessel or non-target vessel is present that requires or has a high probability of requiring PCI within 9 months after the index procedure.
5. Bifurcation lesions with planned or high probability of dual stent implantation*
6. Target lesions located within an arterial or saphenous vein graft or distal to a diseased arterial or saphenous vein graft
7. Heavily tortuous or angulated lesions*
8. Lesions containing large thrombus*
9. Total occlusions*
10. Lesions present within 10mm of another lesion treated by PCI*
11. Restenotic lesions* *Refers to target lesions. Non-target lesions not meeting these criteria may be treated as appropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-08 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
%NIH volume | at 9 months
  NIH volume/stent volume × 100 at 9 months as measured by the OCT core laboratory (all doses pooled vs. placebo).

SECONDARY OUTCOMES:
%NIH at minimum lumen area (MLA) site | 9 months
  Secondary OCT endpoint evaluated at 9 months as measured by the OCT core laboratory
MLA | 9 months
  Secondary OCT endpoint evaluated at 9 months as measured by the OCT core laboratory
% area stenosis | 9 months
  Secondary OCT endpoint evaluated at 9 months as measured by the OCT core laboratory
% stent strut coverage | 9 months
  Secondary OCT endpoint evaluated at 9 months as measured by the OCT core laboratory
In-stent late loss | 9 months
  Secondary angiographic endpoint evaluated at 9 months
In-segment percent diameter stenosis (%DS) (within 5mm margins proximal and distal to stent) | 9 months
  Secondary angiographic endpoint evaluated at 9 months
In-stent %DS | 9 months
  Secondary angiographic endpoint evaluated at 9 months
In-segment late loss | 9 months
  Secondary angiographic endpoint evaluated at 9 months
In-stent late loss compared between the 3 doses of the study drug | 9 months
  Secondary angiographic endpoint evaluated at 9 months
In-segment binary restenosis (stenosis of >50% of the vessel diameter) | 9 months
  Secondary angiographic endpoint evaluated at 9 months
In-stent minimum lumen diameter (MLD) | 9 months
  Secondary angiographic endpoint evaluated at 9 months
Length and patterns of angiographic restenosis (Mehran classification) | 9 months
  Secondary angiographic endpoint evaluated at 9 months
MACE | 30 days, 9 months, 1 year
  Clinical: The composite rate of cardiac death, any MI or ischemia-driven TLR
Clinically driven TLR | 30 days, 9 months, 1 year
  Clinical: Defined as re-intervention (PCI or CABG) due to stenosis of ≥50% at the level of the index-targeted lesion(s) (inside 5mm proximal and distal to the implanted stent), by quantitative coronary angiography (QCA), with ischemic signs and/or symptoms
Clinically driven target vessel revascularization (TVR) | 30 days, 9 months, 1 year
  Clinical: Defined as re-intervention (PCI or CABG) due to stenosis of ≥50% inside the targeted epicardial vessel, by QCA, with ischemic signs and/or symptoms
TVF | 30 days, 9 months, 1 year
  Clinical: Defined as the composite of cardiac death, target vessel MI, or clinically driven TVR
TLF | 30 days, 9 months, 1 year
  Clinical: Defined as the composite of cardiac death, target vessel MI, or clinically driven TLR
Target Vessel Related MI | 30 days, 9 months, 1 year
  Clinical: The number of patients who suffer a MI that is related to the target vessel of the procedure.
Stroke | 30 days, 9 months, 1 year
  Clinical: Major, minor and transient ischemic attack; secondary clinical endpoint evaluated at 30 days, 9 months, and 1 year post procedure
All death | 30 days, 9 months, 1 year
  Clinical: The number of patients who die from all causes
MI | 30 days, 9 months, 1 year
  Clinical: The number of patients who suffer a myocardial infarction
Composite endpoint of cardiac death or MI | 30 days, 9 months, 1 year
  Clinical: The number of patients who die of cardiac-related causes or myocardial infarction
Definite or probable ARC defined stent thrombosis | 30 days, 9 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Généreux, MD, Principal Investigator — Cardiovascular Research Foundation (CRF)
Locations (1):
- Kaplan Medical Center, Rehovot, Israel

REFERENCES:
- [Derived] Genereux P, Chernin G, Assali AR, Peruga JZ, Robinson SD, Schampaert E, Bagur R, Mansour S, Rodes-Cabau J, McEntegart M, Gerber R, L'Allier P, de Silva R, Daneault B, Aggarwal SK, Dzavik V, Ozan MO, Ben-Yehuda O, Maehara A, Stone GW, Jonas M. Double-blind, placebo-controlled evaluation of biorest liposomal alendronate in diabetic patients undergoing PCI: The BLADE-PCI trial. Am Heart J. 2022 Jul;249:45-56. doi: 10.1016/j.ahj.2022.03.004. Epub 2022 Mar 17. PMID 35305955